CLINICAL TRIAL: NCT05939284
Title: Progesterone-Primed Ovarian Stimulation Might be a Safe and Effective Alternative to GnRH-antagonist Protocol for Controlled-Ovarian Stimulation of Infertile PCOS Women
Brief Title: Progesterone-Primed Ovarian Simulation in Controlled-ovarian Simulation of Infertile PCOS Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Walid Mohamed Elnagar, Assistant professor of gynecology, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZU-IRB #10874-25/6-2023
Record Dates: First submitted 2023-07-03; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: PCOS

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group C (Active Comparator)
  Interventions: Drug: Injection of Cetrorelix
- Group S (Active Comparator)
  Interventions: Drug: Oral insertion of dydrogeserone

INTERVENTIONS:
Drug: Injection of Cetrorelix — Patients received Cetrorelix subcutaneous injection on the day-6 in a dose of 0.25 daily till the trigger day.
  Arms: Group C
Drug: Oral insertion of dydrogeserone — Patients received dydrogesterone in an oral dose of 20 mg/day in parallel with gonadotropin injection from day-2 of the menstrual cycle till the trigger day
  Arms: Group S

SUMMARY:
The study evaluated the safety and efficacy of the progesterone-primed ovarian stimulation (PPOS) coupled with gonadotropin (FSH) for infertile women with polycystic ovary syndrome (PCOS) who were assigned for ICSI and frozen blastocyst transfer.

200 infertile women were divided randomly into Group C, which received Cetrorelix injection (0.25 mg daily) on day-6, and Group S, which received oral dydrogesterone (20 mg/day) on day-2 of the menstrual cycle till the trigger day. All patients received an FSH injection of 225 IU daily from day-2 till triggering day. ICSI was performed and day-5 blastocysts underwent vitrification ultra-rapid cryopreservation till being transferred. Outcomes included the ability of PPOS to suppress the premature luteinizing hormone (LH) surge and prevent the development of ovarian hyperstimulation syndrome (OHSS), the incidence of profound LH suppression, the number of retrieved M2 oocyte and fertilization, chemical and clinical pregnancy rates, and the miscarriage rate.

ELIGIBILITY:
Inclusion Criteria:

* Infertile PCOS women;
* aged 20-35 years;
* had BMI <35 kg/m2.

Exclusion Criteria:

* Women who were younger than 20 or older than 35 years,
* obese of grade II or III,
* had poor OR, other causes of infertility,
* had previous attempts of IVF, had a history of repeated pregnancy loss.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 238 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-09-14 (Actual); Study Completion 2023-01-25 (Actual)

PRIMARY OUTCOMES:
Success rate of PPOS in relation to Premature LH surge suppression | 12 months
  the success rate of PPOS as regards the suppression of premature LH surge and prevention of the development of OHSS.

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig university, Zagazig, Ash Sharqia Governorate, Egypt